CLINICAL TRIAL: NCT07130721
Title: Assessment of Blood Biomarkers (D-dimer and C-Reactive Protein) in Predicting Cardiovascular Complications Among Hemodialysis Patients: A Cross-Sectional Study
Brief Title: Assessment of D-dimer and CRP for Cardiovascular Risk Prediction in Hemodialysis Patients
Acronym: BIOCARD-HD
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mennat Allah Mahmoud Ahmed, MSc Candidate, Faculty of Medicine, Assiut University, Assiut University
Other Study IDs: 04-2025-201318
Record Dates: First submitted 2025-08-09; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: End Stage Renal Disease on Dialysis
MeSH Terms: interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemodialysis Patients without Cardiovascular Disease: Patients undergoing regular hemodialysis for at least 3 months with no clinically documented cardiovascular disease. Cardiovascular status is confirmed by reviewing medical records, ECGs, and other relevant reports.
  Interventions: Diagnostic Test: C-Reactive Protein (CRP) Test; Diagnostic Test: D-dimer Test; Diagnostic Test: Electrocardiogram (ECG)
- Hemodialysis Patients with Cardiovascular Disease: Patients undergoing regular hemodialysis for at least 3 months with confirmed cardiovascular disease based on medical records, ECGs, echocardiography, or documented hospital admissions
  Interventions: Diagnostic Test: C-Reactive Protein (CRP) Test; Diagnostic Test: D-dimer Test; Diagnostic Test: Electrocardiogram (ECG)

INTERVENTIONS:
Diagnostic Test: C-Reactive Protein (CRP) Test — Blood samples will be collected once from all participants to measure CRP levels
Diagnostic Test: D-dimer Test — D-dimer levels will be assessed once to evaluate thrombotic risk.
Diagnostic Test: Electrocardiogram (ECG) — A standard 12-lead ECG will be performed once per participant to assess cardiovascular status

SUMMARY:
This study aims to assess whether two blood markers - C-reactive protein (CRP) and D-dimer - can help predict cardiovascular complications in patients undergoing regular hemodialysis. Cardiovascular disease is a common and serious problem in dialysis patients, and early detection is important.

the study will include 100 adult patients from the Hemodialysis Unit at Assiut University Hospital. Participants will be divided into two groups: those with and those without known heart disease. Each participant will have a one-time blood test to measure CRP and D-dimer levels. In addition, an electrocardiogram (ECG) will be done once to check for signs of heart problems.

DETAILED DESCRIPTION:
This cross-sectional study is designed to explore the potential role of hematologic biomarkers in predicting cardiovascular complications among patients undergoing maintenance hemodialysis. Cardiovascular disease is a leading cause of morbidity and mortality in this population, and systemic inflammation and hypercoagulability are thought to contribute significantly to adverse outcomes.

C-reactive protein (CRP) is a well-established marker of systemic inflammation, while D-dimer reflects activation of the coagulation and fibrinolytic pathways. Both biomarkers have been associated with increased cardiovascular risk in the general population, but their predictive value in hemodialysis patients remains insufficiently characterized.

A total of 100 adult patients on maintenance hemodialysis will be evaluated. The population will be stratified into two groups based on the presence or absence of clinically confirmed cardiovascular disease. Laboratory analysis will include measurement of CRP and D-dimer, and cardiovascular assessment will include a standard 12-lead ECG. Clinical and demographic data will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years

On regular hemodialysis for at least 3 months

Able and willing to provide informed consent

Group I: Hemodialysis patients with no clinically documented cardiovascular disease

Group II: Hemodialysis patients with confirmed cardiovascular disease (by medical records, ECGs, echocardiography, or documented hospital admissions)

Exclusion Criteria:

* Acute or recent infection (within the past 4 weeks)

Use of anticoagulant or antiplatelet therapy

Active malignancy

Autoimmune or chronic inflammatory disease

Known bleeding or thrombotic disorders

Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients treated at the Hemodialysis Unit of Assiut University Hospital, including those with and without documented cardiovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Serum CRP level among hemodialysis patients | At baseline (one-time measurement)
  To assess the level of serum CRP in hemodialysis patients with and without cardiovascular disease and compare values between the two groups to explore possible associations
Plasma D-dimer level among hemodialysis patients | At baseline (one-time measurement)
  To assess the level of plasma D-dimer in hemodialysis patients with and without cardiovascular disease and compare values between the two groups to explore possible associations.

SECONDARY OUTCOMES:
Presence of cardiovascular abnormalities on ECG | At baseline (one-time measurement)
  To assess cardiovascular status of hemodialysis patients using a standard 12-lead ECG and record the presence of abnormal findings

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because the study involves sensitive health data and patient confidentiality must be maintained.